CLINICAL TRIAL: NCT03741439
Title: Randomized Controlled Trial to Test Low Intensity Shockwave Treatment in Patients With Mild and Moderate Erectile Dysfunction Using a Electromagnetic Emitter
Brief Title: RCTrial to Test Low Intensity Shockwave Treatment in Patients With Mild/Moderate Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IVI Santiago de Chile (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other); University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Marconi01
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Erectile Dysfunction; Endothelial Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and who analyzes the data are blind to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Receives real treatment according to manufactures instructions. 6 sessions of low intensity shockwave treatment with an electromagnetic emitter.
  Interventions: Device: Treatment
- Sham Arm (Sham Comparator): Receives sham treatment with same applicator, same sound, same time and number of shocks. But no real energy is delivered.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Treatment — Low intensity shockwave treatment in patients with mild/moderate ED using a electromagnetic emitter
  Arms: Treatment arm
Device: Sham — Sham treatment
  Arms: Sham Arm

SUMMARY:
Even though, the efficacy of Low-Intensity Shockwave Therapy (LIST) to treat Erectile Dysfunction (ED) has been documented by numerous trials; it is still not recommended by clinical guidelines. Different types of: shockwave generators, treatment protocols and ED severities of patients included in the studies, explain the lack of recommendations for a standard treatment. Ideally, each shockwave generator should have its own efficacy data from randomized controlled trials, using standardized protocols, and in defined populations.

Objective: to test the efficacy of a electromagnetic shockwave generator (Dornier Aries) in treating patients with mild and moderate ED in a randomized controlled trial.

Patients and methods: 38 patients with mild/moderate ED (IIEF-5= 11-21), are being prospectively randomized (1:1) to receive 6 sessions of LIST or sham (same: number of sessions, time and sound, with out transmitting energy). The patients and who analyzed the data are blind to randomization. The following parameters were analyzed: IIEF-5, IIEF-15, Sexual Encounter Profile (SEP) 2 and 3, Global Assessment Question (GAQ) 1 and Erection Hardness Score (EHS) at: baseline (T0), at the end of the 6 sessions (T1); at 6 (T2) and 12 weeks (T3). During all the study patients were instructed to receive no other treatment for ED.

After ending T3 we expect to treat placebo patients to see impact of changing arm study.

DETAILED DESCRIPTION:
We are test the efficacy of a electromagnetic shockwave generator (Dornier Aries) in treating patients with mild and moderate ED in a randomized controlled trial.

Patients and methods: 38 patients with mild/moderate ED (IIEF-5= 11-21), are being prospectively randomized (1:1) to receive 6 sessions of LIST or sham (same: number of sessions, time and sound, with out transmitting energy). The patients and who analyzed the data are blind to randomization. The following parameters were analyzed: IIEF-5, IIEF-15, Sexual Encounter Profile (SEP) 2 and 3, Global Assessment Question (GAQ) 1 and Erection Hardness Score (EHS) at: baseline (T0), at the end of the 6 sessions (T1); at 6 (T2) and 12 weeks (T3). During all the study patients were instructed to receive no other treatment for ED.

After ending T3 we expect to treat placebo patients to see impact of changing arm study.

ELIGIBILITY:
Inclusion Criteria:

* Mild/moderate erectile dysfunction
* Good response to any phospodiesterase inhibitor

Exclusion Criteria:

* No history of erectile dysfunction
* No decompensated diabetes
* No untreated hypogonadism
* No severe erectile dysfunction

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men because is for erectile dysfunction.
Enrollment: 38 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-01-02 (Estimated)

PRIMARY OUTCOMES:
Changes in IIEF-5 | 12 weeks
  We expect a change of 3.5 points in the IIEF-5 score

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Marconi, MD, Principal Investigator — Asistant Professor Urology Department Universidad Catolica de Chile
Locations (1):
- Unidad de Andrologia - Red Salud UC/Christus, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
We are evaluating is we decide to share all the protocol. All the protocol will be published with the results.